CLINICAL TRIAL: NCT01323868
Title: Endogenous Endophthalmitis Rates, Clinical Course, and Outcomes
Brief Title: Endogenous Endophthalmitis in the Inpatient Setting
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theodore Leng, Clinical Assistant Professor of Ophthalmology, Stanford University
Other Study IDs: SU-03232011-7621; IRB-18785
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the rate of endogenous endophthalmitis in patients admitted to Stanford Hospital with a systemic infection and positive blood cultures, as this may improve the clinical care of this population of patients.

DETAILED DESCRIPTION:
Some patients admitted to the hospital have blood-borne infections. Occasionally, these blood infections can end up inside the eye and cause an infection inside the eye (called endogenous endophthalmitis).

Prior to modern and rapid treatment of systemic infections, the rate of endogenous endophthalmitis was reported to be 37% in 1982. By 1997, the rate was reported to be 2.8%. This study aims to determine the rate of endogenous endophthalmitis at Stanford Hospital in the modern medical era in that our rates may be different as those reported in the literature. This potential difference may be a reflection of treatment protocols and antibiotics currently in use at Stanford Hospital.

ELIGIBILITY:
Inclusion Criteria:All patients admitted to Stanford Hospital that have a systemic blood-borne infection and on which an Ophthalmology consult to rule out endogenous endophthalmitis is performed will be included in the study. Exclusion Criteria:None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients at Stanford Hospital with positive blood cultures who receive an Ophthalmology consultation and eye examination.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Positive intraocular infection | 1 day

SECONDARY OUTCOMES:
Visual acuity | 2 wk

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Leng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States